CLINICAL TRIAL: NCT04003948
Title: Preliminar Efficacy and Safety of Ibogaine in the Treatment of Methadone
Brief Title: Preliminary Efficacy and Safety of Ibogaine in the Treatment of Methadone Detoxification
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Center for Ethnobotanical Education, Research, and Service (Other)
Collaborators: Multidisciplinary Association for Psychedelic Studies (Other); University Rovira i Virgili (Other); Universidad Autonoma de Madrid (Other); Hospital Universitari Sant Joan de Reus (Other); University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IBO-METAD-001
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Drug Dependence; Drug Use Disorders; Opioid Dependence
Keywords: Ibogaine; Methadone; Drug dependence; Addiction
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed dose (Experimental): Ibogaine Hydrochloride 100 mg on each administration.
  Interventions: Drug: Ibogaine Hydrochloride
- Ascending dose (Experimental): Ibogaine Hydrochloride on ascending doses (100-200-300-400-500-600).
  Interventions: Drug: Ibogaine Hydrochloride

INTERVENTIONS:
Drug: Ibogaine Hydrochloride — Fixed or ascending doses of ibogaine will be administered for the treatment of opioid withdrawal syndrome.

SUMMARY:
Methadone is a very long-acting opiate very difficult to detox from. In Spain there are a lot of methadone dependent people in the aftermath of the heroin epidemic of the 1980s. Many have been dependent for more than 15 years and a number of them have a relatively stable life condition (have work, family, housing, etc.) and a relatively good health condition in comparison with current heroin users. This Phase-II RCT is a collaboration with the Sant Joan Hospital in Reus, Spain. Twenty patients on the methadone maintenance program will be recruited. Patients will be randomized to two groups: One receiving 6 doses of 100 mg of ibogaine; and the other one receiving ascending doses of ibogaine (100-200-300-400-500-600). Methadone use will be interrupted and for both groups ibogaine will be administered when clinical symptoms of opioid withdrawal appear. After an ibogaine dose, when symptoms of opioid withdrawal appear again, half of the methadone dose used last time will be administered. By doing so, methadone doses will be progressively reduced until no withdrawal symptoms appear.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years.
* Body weight within normal range (Quetelet's index between 19 and 27) expressed as weight (kg) / height (m2).
* Normal clinical records and physical examination.
* Subjects without organic disorders.
* Laboratory tests (hematology, biochemistry and urinalysis) within the range of normal values, according to the laboratory reference values of the "Hospital Universitari Sant Joan de Reus". Variations may be admitted according to the clinical criteria of the Principal Investigator.
* Clinically acceptable temperature, blood pressure and pulse rate in supine and standing position (SBP between 100-140 mm Hg/ DBP between 50-90 mm Hg / HR between 50-100 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
* Having not participated in another clinical trial in the last 2 months.
* Free acceptance to participate in the study by obtains signed informed consent form approved by the ethics committee.
* ECG values within the range of normal values (PR < 240 ms, QRS < 110 ms and QTc < 430 ms in men and QTc < 450 ms in women, and heart rate >50 bpm.

Exclusion Criteria:

* Background of allergy, idiosyncrasy or hypersensitivity to drugs..
* Intake of any medication within 2 weeks prior taking the study treatment (except for use of paracetamol in short-term symptomatic treatments), including over-the-counter products (including natural food supplements, vitamins and medicinal plants products), or any enzymatic inductor or inhibitor before the drug administration.
* Viral activity for hepatitis B, C or HIV.
* Background or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological or neurological disease or other chronic diseases.
* History of severe psychiatric disease like psychosis, bipolar disorder or dissociative disorders, or a high risk to develop them as reported by psychometric questionnaires.
* Past or current risk of suicide.
* Having undergone major surgery during the previous 6 months before the enrollment.
* Positive results of the drugs at screening period or the day before starting treatment period: Amphetamines, Cocaine, Ethanol, Opiates (not methadone), and not prescribed Benzodiazepines (positive results may be repeated at the discretion of the PI).
* Not understanding the nature of the study and potential consequences.
* 12 lead ECG obtained at screening with PR ≥ 220 msec, QRS ≥120 msec and QTc ≥ 440 msec for men and ≥450 for women, bradycardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval.
* Pregnancy or lactation status (females).
* Not understanding the informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Methadone dose | 0-6 months
  Rate of decrease of methadone dose used

SECONDARY OUTCOMES:
Adverse events | 0-24 hours
  Description of adverse events found at different doses of ibogaine
Cardiovascular effects | 0-24 hours
  Electrocardiogram (QT interval, ST wave)

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos Bouso, PhD, Principal Investigator — International Center for Ethnobotanical Education, Research, and Service; Tre Borràs, MD, Principal Investigator — Hospital Universitari Sant Joan de Reus; Genís Ona, MSc, Study Director — International Center for Ethnobotanical Education, Research, and Service
Locations (1):
- Hospital Universitari Sant Joan, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No